CLINICAL TRIAL: NCT03287128
Title: A Retrospective Analysis of the Outcome of Patients With Relapsed/Refractory Acute Myeloid Leukemia (AML) Included in a Patient Named Program of Gemtuzumab Ozogamicin/Mylotarg®
Brief Title: Retrospective Analysis of the Outcome of Patients With Relapsed/Refractory Acute Myeloid Leukemia Included in a Patient Named Program of Gemtuzumab Ozogamicin/Mylotarg®
Acronym: MYLOR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, Ms Juliette LAMBERT, study Coordinator, Versailles Hospital
Other Study IDs: P1612_MYLOR
Record Dates: First submitted 2017-09-15; First posted 2017-09-19 (Actual); Last update posted 2018-01-24 (Actual); Status verified 2017-09

CONDITIONS: Leukemia, Myeloid, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Gemtuzumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Gemtuzumab Ozogamicin (GO) — patients included in a compassionate patient named program with GO

SUMMARY:
Gemtuzumab Ozogamicin/Mylotarg® (GO) is a conjugate of a derivative of calicheamicin a potent antitumor anthracycline antibiotic linked to a recombinant humanized antibody against the CD33 antigen. Pivotal phase 2 study in relapsed AML adult patients used GO 9 mg/m2 as a monotherapy on days 1 and 14, and showed a 30% response rate with half CR and CRp (CR with incomplete platelets recovery). Four randomized studies, 3 in adults and 1 in children, performed in patients with non-previously treated AML tested the addition of lower doses of GO ( 3mg or 6 mg/m2) to standard induction chemotherapy and showed benefit on survival endpoints. Results from these studies were available in 2011 in adults and 2014 in children. In 2010 the french health agency (ANSM) opened a compassionate patient named program (authorization for temporary utilization (ATU) program) of GO in relapsed/refractory AML patients. Patients were orally informed about the status of the GO. From 2010 to 2012 it was recommended to use GO as a monotherapy at a dose of 9mg/m2 on days 1 and 14 according to the protocol used in pivotal phase 2 study. After 2012 it was recommended by the health authority to use GO at the dose of 3 or 6 mg/m2 in addition to chemotherapy regarding the toxicity of higher dose given once.

From 2010 to 2015 more than 500 AML patients have been included in this ATU program.

The main objective of the study presented here is to assess the efficacy and safety of GO 3 or 6 mg/m2 (single dose or fractionated GO) given in as treatment of relapsed/refractory AML in adult patients.

The coordinator choose to collect the data from centers that included 10 patients or more from January 2012 to December 2015.

This represents approximately 420 patients from 33 hematology departments.

ELIGIBILITY:
Inclusion Criteria:

* Patient more than 18 year old;
* De novo or secondary leukemia.
* Refractory to standard intensive chemotherapy (defined by the association of anthracycline and cytarabine, at different doses) or in first relapse.
* Treated with GO from January 2012 to December 2016.

Exclusion Criteria:

* Previous treatment with GO
* AML type 3
* More than 1 relapse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective cohort, using medical charts of relapsing or refractory patients after intensive chemotherapy included in a compassionate patient named program of Gemtuzumab Ozogamicin from January 2012 to December 2015 and treated in 30 centers to evaluate the efficacy and safety of Gemtuzumab Ozogamicin (GO) given in addition to chemotherapy.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-10-01 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
Remission rate including complete remission (CR) and complete remission with incomplete hematological recovery (CRi). | 45 days

SECONDARY OUTCOMES:
Overall survival defined as the time from onset of GO re-treatment for relapsed/refractory AML to the date of death. | 2 years
Duration of second remission | 2 years
Relapse Free Survival defined as the time from onset of GO retreatment for relapsed/refractory AML to the first event (death or relapse). | 2 years
Cumulative incidence of early deaths | 60 days
Grade 3 to 5 liver, infectious and cardiac adverse events | 45 days
Severe adverse events during induction treatment | 45 days
Cumulative incidence of allogenic transplant among responder's patients with respects to age. | 2 years

CONTACTS AND LOCATIONS:
Locations (11):
- France (11):
  - C.H.U. d'Amiens - Hôpital Sud, Amiens
  - C.H.U. d'Angers, Angers
  - HIA Percy, Clamart
  - Hôpital Henri Mondor, Créteil
  - Hôpital du Bocage, Dijon
  - Hôpital André Mignot, Le Chesnay
  - Hôpital Hotel Dieu, Nantes
  - Hôpital de la Source, Orléans
  - Hopital Saint Louis, Paris
  - C.H. Lyon Sud, Pierre-Bénite
  - Hôpital Brabois Adultes, Vandœuvre-lès-Nancy